CLINICAL TRIAL: NCT04348942
Title: COVID-19 Study - A Primarily Prospective Observational Study of COVID-19 Clinical Characteristics and Acquired Immune Response Within the General Population
Brief Title: A COVID-19 Symptom, Exposure and Immune Response Registry
Status: Completed | Type: Observational
Sponsor: ObvioHealth (Industry)
Responsible Party: Sponsor
Other Study IDs: OBVIO-OBV-001
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a 6-month, 100% remote study that will collect a broad range of data that may provide insight into the COVID-19 global pandemic. Data collected will include participant medical histories, history of prior SARS-CoV-2 infection and exposure to known cases. On an ongoing basis data will be collected on new contacts with known cases, the presence of COVID-19 symptoms, including severity and outcome, and information on the immune system response to SARS-CoV-2 infection.

DETAILED DESCRIPTION:
This is a 6-month, 100% remote study that will collect a broad range of data that may provide insight into the COVID-19 global pandemic. All data will be collected by participant entry into a mobile app designed for this study.

Upon entering the study, participants will be asked a series of questions about their prior exposure to the SARS-CoV-2 virus including reporting prior test results, and identification and description of contact with known or cases or other high risk encounters. Participants will also provide a detailed medical history.

On on ongoing basis, participants will be asked to report any symptoms associated with COVID-19 that they develop, and any new contacts they experience with known cases. Some participants will be sent an at-home SARS-CoV-2 antibody test and asked to report the results. In addition, participants will be asked to report the result of any other test they receive for COVID-19 outside of the study.

ELIGIBILITY:
Inclusion Criteria:

* Open to any adult individuals (18 years of age or older) permanently residing in the United States
* Have regular access to smartphone and internet sufficient to support registry demands
* Willing and able to follow the procedures of the study
* Willing and able to provide informed consent

Exclusion Criteria:

* Participants unable to understand the study protocol or provide informed consent
* Participants unable or unwilling to perform all requested study tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults residing in the USA, regardless of past or current COVID-19 status
Sampling Method: Non-Probability Sample
Enrollment: 804 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-21 (Actual)

PRIMARY OUTCOMES:
Registry Data | 6 months
  Compilation of registry data via regular self-reported questionnaires on symptoms (known to be associated with COVID-19 diagnosis including presence, severity, and duration using the Obvio-19 app.

CONTACTS AND LOCATIONS:
Locations (1):
- ObvioHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah P, Magee K, Buccellato KH, Ismond M, Watson J. Real world data on cardiometabolic diseases in U.S. adults during the SARS-CoV-2 pandemic: a decentralized registry study. Cardiovasc Diabetol. 2022 Feb 14;21(1):24. doi: 10.1186/s12933-022-01462-3. PMID 35164745